CSMC Date Effective: 4/7/2023



## ASSENT FOR TEENS 13-17 YEARS OF AGE / PARENTAL PERMISSION\* / CONSENT FORM FOR RESEARCH

\*This form will also serve as a Permission Form for your child to participate in this research. In this case, "You" refers to "Your child" and "you"

**Title:** Transcending COVID-19 barriers to pain care in rural America: Pragmatic comparative effectiveness trial of evidence-based, on-demand, digital behavioral treatments for chronic pain

**SPONSOR:** THE NATIONAL INSTITUTES OF HEALTH (NIH)

PRINCIPAL INVESTIGATOR: BRENNAN SPIEGEL, MD, MSHS

STUDY CONTACT PHONE NUMBERAT CSMC: (310) 423-0684

**AFTER HOURS CONTACT (24 HOURS):** (248) 383-5346

This research study is sponsored by the NIH. The NIH only reimburses Cedars-Sinai Medical Center for the costs associated with running the study; the NIH is not providing additional compensation to Cedars-Sinai Medical Center or the Principal Investigator for their participation in the study.

## **KEY INFORMATION ABOUT THIS RESEARCH STUDY**

We are seeking your consent to take part in this research study. Your participation in this research is voluntary. If you choose to participate, you can stop at any time. Please consider the following summary, along with the more detailed information provided throughout this consent form.

- The purpose of this study is to compare the impact of painTRAINER® with virtual reality (VR) therapy on chronic pain. We want to see which treatment will more effectively improve pain management, offer additional pain relief, or be an effective alternative to traditional pain medication.
- The main procedures of this study include using a mobile health application or a virtual reality headset every day to manage your pain for 60 days. If you are provided the virtual reality headset, using the device will take about 10 minutes each day. We will also ask you to complete weekly surveys over the first 30 days, then biweekly surveys until the end of the study. Surveys will be sent via email and can be

CSMC Date Effective: 4/7/2023

completed from a computer or smartphone (Android or iOS). You will need to complete one week of screening surveys prior to being given access to the mobile health application or being sent the virtual reality headset and other study materials. If assigned to the VR group, the virtual reality headset will be provided to you for the duration of the study at no cost. If you choose to take part in this study, it will last about 60 days.

- All research studies involve some risks. Risks or discomforts from this study may include: minor psychological distress from questionnaires regarding health and employment status, risk of neck pain from wearing the headset, and ~5% risk of "cybersickness," presenting as short-term symptoms related to entering VR environments (vertigo, nausea, headache).
- Potential immediate benefits include reduction of chronic pain and overall improvements in psychological health. Potential long-term benefits include improved functionality, reduced opioid use, and improvements in overall physical health. This research will contribute to the societal knowledge about the use of digital interventions within healthcare.
- If at any point in the study you feel the need to make any changes to your prescribed medications, please talk with your prescribing physician. Making abrupt changes to medications may be unsafe and any modification in medications should occur under the guidance of your physician.
- If you choose not to participate, there may be other choices available to you. You can continue your current treatment with your providers. You will not lose any services, benefits or rights you would normally have if you choose not to participate. Please discuss your choices with the researchers.

Please take time to read this entire form and ask questions before deciding whether to participate in this study. You are encouraged to talk with family members, friends, and/or healthcare providers before you make your decision.

## 1. WHAT IS THE PURPOSE OF THIS RESEARCH STUDY?

This study will compare two available, evidence-based, digital pain treatment programs that patients can use at home. The goal is to see if one approach is better than the other, and whether certain patients respond to one more than the other. We want to know if the use of this tool can limit the extent to which pain interferes with your life and if your overall health improves.

You are being asked to take part in this research study because you are a patient at either Cedars-Sinai Medical Center, Ochsner Health, UAB Medicine, or BendCare Physician network and have chronic pain.

In this study, two available, evidence-based, digital pain treatment programs will be assessed for their ability to reduce pain. You will be randomized into one of two groups after the

CSMC Date Effective: 4/7/2023

screening period. See Section 2 below for more information.

The study will enroll up to 300 people in total.

This research study is designed to use painTRAINER®. painTRAINER® is among the most widely-validated mHealth interventions for pain management. The app teaches evidence-based pain coping skills using a self-administered, home-based software program. The system delivers eight sessions via any web-connected platform, including Android or iOS smartphones, tablets, or personal computers. The digital curriculum covers progressive muscle relaxation, activity/rest cycling, pleasant activity scheduling, recognizing negative automatic thoughts, pleasant imagery/distraction, problem solving, and monitoring for maintenance. Patients complete one session per week in a pre-determined order. The program can be completed in a flexible manner to accommodate life and medical events.

This research study is also designed to use the PICO G2 Headsets. The VR headset are not currently regulated by the FDA and pose minimal to no risks to individuals.

## 2. WHAT WILL HAPPEN DURING THE STUDY?

This section provides a general overview of what will happen during your participation in this study. Information included below should be considered along with the flowchart of procedures attached as an Appendix.

The flowchart shows a timeline for research-related procedures that are involved in your participation in this study. **Research-related procedures** are those performed solely for the research. They would not be performed if you did not take part in the study. All procedures in this study are research-related procedures.

At the start of the study, you will be sent surveys via email. Surveys can be completed on a computer or smartphone (Android or iOS). You will be trained on how to use painTRAINER®, or the VR headset and any related apps required for the study.

#### Overview of study:

This is a randomized research study with an additional screening week. Standard (routine) care will involve treatment as prescribed by your provider for your pain condition. Your study participation will not dictate your standard treatment or care.

- "Randomized" means that you will be assigned to a study group by chance, like flipping a coin. You will be randomized into one of the two study groups and will have an equal chance of being placed in each group below.
- "Screening week" means you will receive surveys every day for a week via email. Once you complete this week of surveys, you will be eligible to be randomized.



CSMC Date Effective: 4/7/2023

A computer will randomly assign you to a study group. This is done because no one knows if the results experienced by the participants in one study group are better, the same, or worse than the results experienced by participants in the other. Once you are put in one group, you cannot switch to another group. Neither you nor your doctor can choose the group in which you will be placed.

Any of these different approaches could help your condition but could also cause mild temporary side effects. This study will allow the researchers to learn whether the different software programs are better, the same, or worse than the current standard of care. Audiovisual therapy and mobile health application have been used in several studies at Cedars-Sinai. The results of these studies have demonstrated the device to be safe; less than 25% of patients who use the VR headset have minor, short-term side effects from the device.

If you are assigned to any group, you will be followed as you receive the care generally provided for individuals with your condition. You will either be asked to use the VR unit for no more than 20 minutes at least once a day and as needed during moments of pain or to use painTRAINER® to complete a 35-45 minute session each week. You will be asked to complete surveys asking questions about your pain via email.

The VR unit, and the app we install on your smartphone will collect data and periodically upload data to secure, encrypted servers at Cedars-Sinai.

You will be asked to keep your smartphone on your person and answer surveys when prompted. We will also ask you to keep the VR headset with you whenever possible. In the event that any of the study equipment are lost or damaged, you will not be held responsible for the lost or damaged study equipment. However, all study equipment, whether damaged or intact, must be returned at the end of the study.

## Prescription Data

As part of this study, we will be collecting prescription data from the Cedars-Sinai Medical Record.

## How long will you be in the study?

We think you will be in this study for about 60 days.

## 3. WHAT ARE THE POSSIBLE RISKS?

This section describes the possible risks and/or discomforts we anticipate you could experience that are related to the study procedures:

#### VR Intervention:

While using the VR headset, you may experience discomfort with the virtual environment, including temporary headache, vertigo, or nausea. These should be short-term and should stop soon after the headset is removed. You may also experience neck pain if using the headset.

You may use glasses with the VR headset. With proper usage, the headset will not damage

CSMC Date Effective: 4/7/2023

your glasses. Please follow usage instructions as the research team is not responsible for any damage to glasses that may occur from misuse of the equipment.

## Surveys:

It is possible that some of the items in the surveys may make you feel uncomfortable or embarrassed. You are not required to respond to any item that you do not wish to answer. The surveys will be labeled with a unique study number that will link your identity so that only the research team can recognize you.

There are no anticipated long-term risks from participating in this study and no short term risk for using the painTRAINER®.

#### Risks of sharing data

Even though we will protect your privacy as much as possible, there is a very small chance that the data could be identified as yours. The risk of this happening is very small, but may increase in the future as technology changes.

Research using data from this study may lead to new tests, drugs, or devices with commercial value. You will not receive any payment for any product developed from research using your samples and data.

If you do not want your data and samples used for other research, you should not participate in this study.

#### Follow-up Visit for Discontinuing Participants

While you are free to discontinue your participation at any time, we encourage you to complete the final study questionnaire on the  $60^{th}$  day.

## 4. ARE THERE BENEFITS IN TAKING PART IN THE STUDY?

If you agree to take part in this research study, there may or may not be direct medical benefit. The possible benefits of taking part in the research study are pain relief, improved functionality, greater satisfaction with care, and overall improvements in physical and mental health. However, no benefit is guaranteed. It is possible that your condition may remain unchanged or even get worse.

It is possible that none of the programs we are testing will provide benefit. However, you will continue to receive standard of care treatment from you physician regardless of the group you are assigned to. Your participation will also help us by advancing scientific knowledge about pain management.

We hope the information learned from this research study will benefit other individuals with pain in the future by helping us to learn how we can reduce pain and improve functionality, while minimizing the use of opioids.

## Potential benefits of sharing of data

There is no direct benefit to you from the storage and sharing of your data, but sharing may

CSMC Date Effective: 4/7/2023

help researchers learn more about pain management, which may help you or others in the future.

## 5. WHY WOULD MY PARTICIPATION BE STOPPED?

Your participation in this study may be stopped at any time by the researcher or the sponsor without your consent for any reason, including:

- The study is stopped or suspended;
- Funding for the study is reduced, stopped or withdrawn;
- If it is in your best interest;
- You do not consent to continue in the study after being told of changes in the research that may affect you;
- You do not follow the study procedures.

You may choose (or you may be required) to withdraw from certain parts of the study, but invited to continue with other parts. For example, you might stop using the audiovisual experience, but continue to fill out the surveys. Separate written consent will be requested if your continued participation will involve procedures not described in this consent form.

## 6. ARE THERE ANY OTHER OPTIONS?

Your participation is voluntary so you have the right to decline to participate or to withdraw from this research study at any time without any penalty or loss of benefits to which you would be entitled outside of the study. Choosing not to participate will not affect the care you receive at Cedars-Sinai Health System.

## 7. <u>WILL MY INFORMATION BE KEPT CONFIDENTIAL?</u>

We will do our best to make sure that the personal information collected as part of this study is kept private. However, we cannot guarantee total privacy. A copy of your research consent and authorization forms may be filed in your electronic medical record at CSMC. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other identifiable personal information will not be used. Organizations that may look at and/or copy your medical records for research oversight, quality assurance, and data analysis include: accrediting agencies, government and regulatory groups (such as Food and Drug Administration (FDA), Office for Human Research Protections (OHRP), etc.), safety monitors, companies that sponsor the study, and authorized representatives of the sponsor.

Attached to this consent form is an "Authorization Form" that outlines with whom your information may be shared for the purposes of this research and under what circumstances.

We might share your information and/or research samples collected in this study with other researchers at Cedars-Sinai, other academic institutions, or third-party commercial entities for future research without additional informed consent from you. Information that identifies you will be removed and will not be shared with other researchers or anyone outside of Cedars-Sinai.

CSMC Date Effective: 4/7/2023

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Website at any time.

The study will be registered approximately 3 weeks after the first participant is/was enrolled and results will be submitted approximately one year from study completion.

## <u>Protections from Forced Disclosures (Subpoenas) – Certificates of Confidentiality</u>

To further protect your private identifiable information, we have obtained a Certificate of Confidentiality (Certificate) from the federal government.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law such as child abuse and neglect, or harm to self or others.

The Certificate of Confidentiality will not be used to prevent disclosure for any purpose you have consented to in this informed consent document such as including research data in the medical record.

#### **Data Storage and Sharing**

Your study data will be stored securely at Cedars-Sinai. Your data will be stored for 5 years. We will do our best to protect your personal information.

# 8. WHAT IF I BECOME ILL OR INJURED BECAUSE OF TAKING PART IN THIS STUDY?

You will not be in danger of any illness or injury from this research study. However, should

CSMC Date Effective: 4/7/2023

you believe that you are ill or have been injured as a result of your participation, please contact the study team at the phone number listed on page 1 of this consent form.

## 9. <u>FINANCIAL CONSIDERATIONS</u>

#### Costs of Participation

You and your insurance company will not be charged for your participation in this research study. If you choose to receive survey invitations or reminders by text message, your phone number will be shared with Twilio, Inc. If you have a phone plan that includes charges for receipt of text messages, this may result in additional charges on your phone plan. The Sponsor will cover the cost of all items, drugs and services required by this study, including any procedures required by the study that may be standard of care.

## Compensation for Participating

You will be eligible for up to \$300 in Amazon gift card codes at the end of the study. You will be emailed surveys throughout the course of the study. Each email will have a link to a set of surveys:

- After completing 4 of the 5 sets of surveys (80%) in the 1<sup>st</sup> month, you will be sent a \$50 Amazon gift code.
- After you complete 8 of the 10 sets of surveys (80%) in the 2<sup>nd</sup> month and return the equipment, you will be sent a \$225 Amazon gift code. (Participants who receive a VR headset for the duration of the study must return the device in order to receive the \$225 Amazon gift code.)
- Once you complete the week 12 survey, you will be sent a \$25 Amazon gift code

For tax purposes for providing gift card, Cedars-Sinai must collect your name, phone number, address, and the last 4 digits of your Social Security Number. This information will be collected by the research team, but the study team will not keep this information. They will provide it to the Cedars-Sinai financial office for their tax records.

## Financial Interest in the Research

The PI and institution have no potential financial conflict of interest with respect to this study.

## 10. WHAT IF I HAVE QUESTIONS OR PROBLEMS?

Please contact the investigator listed on the first page of this form for questions or concerns about the research.

If you have questions, problems, or concerns that you want to discuss with someone who is not associated with this study, or want to offer suggestions or feedback, please contact:

Cedars-Sinai Human Research Protection Program (HRPP)

Phone: (310) 423-3783

Email: ResearchConcerns@cshs.org

The Cedars-Sinai HRPP has been established to protect the rights and welfare of research

CSMC IRB No: STUDY00001262 / MOD00007536 CSMC Date Effective: 4/7/2023

participants. You may also contact the Cedars-Sinai HRPP if you want to offer input or obtain information regarding the study.

CSMC Date Effective: 4/7/2023

## 11. <u>CONSENT PROVISIONS</u>

If you sign this form below, it means that:

- (1) You have taken the time to carefully read and understand the information presented in this informed consent form; you should discuss it with others, and if appropriate seek a second opinion to make an informed decision;
- (2) The information concerning the research study and its involved procedures has been fully explained to you and your questions have been answered to your satisfaction;
- (3) You have received and understand all of the information you desire regarding your participation in the research study;
- (4) You have considered the potential risks, any anticipated benefits and alternatives (and their relative risks and benefits) of participation;
- (5) You are voluntarily agreeing to participate in this research study;
- (6) You understand that by consenting to participate in the research, you are not giving up any of your legal rights;
- (7) You understand that you have the right to be informed of significant new findings related to this research study which may affect your willingness to continue participating in this study; and
- (8) You have been provided with a copy of the "Experimental Subject's Bill of Rights", if applicable to this research study, and have been provided with an opportunity to ask questions regarding the Bill of Rights.

We will give you a copy of this signed and dated consent form and the Experimental Subject's Bill of Rights.

CSMC IRB No: STUDY00001262 / MOD00007536 CSMC Date Effective: 4/7/2023

## **SIGNATURE PAGE**

## **Consent Form for Research**

**SIGNATURE BY THE PARTICIPANT:** I hereby agree to participate in the research study described to me during the informed consent process and described in this informed consent form. You will be given a signed copy of this form.

| Name of Participant (Print) | ne of Participant (Print) Signature | |
|---|---|---|
| GNATURE BY THE PARTICIPANT'S PARENT/GUARDIAN (If applicable) | | |
| By providing my signature below, I give permission for the participation of my child,, in the research study described in this document. | | |
| Parent/Guardian Name (Print) | Signature | Date of Signature |
| SIGNATURE BY THE INVEST consent described in this form have participant. I further attest that all best of my knowledge. | ve been discussed fully in non-te | echnical terms with the |
| Name of Investigator (Print) | Signature | Date Signed |

CSMC Date Effective: 4/7/2023



#### APPENDIX: EXPERIMENTAL SUBJECT'S BILL OF RIGHTS

In accordance with California Health and Safety Code 24172, any person who is required to consent to participate as a subject in a research study involving a medical experiment or who is requested to consent on behalf of another has the right to:

- 1. Be informed of the nature and purpose of the experiment.
- 2. Be given an explanation of the procedures to be followed in the medical experiment, and any drug or device to be utilized.
- 3. Be given a description of any attendant discomforts and risks to the subject reasonably to be expected from the experiment.
- 4. Be given an explanation of any benefits to the subject reasonably to be expected from the experiment, if applicable.
- 5. Be given a disclosure of any appropriate alternative procedures, drugs or devices that might be advantageous to the subject, and their relative risks and benefits.
- 6. Be informed of the avenues of medical treatment, if any, available to the subject after the experiment if complications should arise.
- 7. Be given an opportunity to ask any questions concerning the experiment or the procedure involved.
- 8. Be instructed that consent to participate in the medical experiment may be withdrawn at any time and the subject may discontinue participation in the medical experiment without prejudice.
- 9. Be given a copy of any signed and dated written consent form used in relation to the experiment.
- 10. Be given the opportunity to decide to consent or not to consent to a medical experiment without the intervention of any element of force, fraud, deceit, duress, coercion, or undue influence on the subject's decision.

CSMC IRB No: STUDY00001262 / MOD00007536 CSMC Date Effective: 4/7/2023

## **APPENDIX: FLOWCHART OF PROCEDURES**

| Procedures | Baseline/<br>Screening | Day 1<br>of<br>Week<br>1 | 8-Week Intervention | | | | | | | Post<br>Intervention | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | 0 | 1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 12 |
| Prospective patients identified (Cohort Builder or Provider) | Х | | | | | | | | | | | |
| Informed consent in person or over phone | X | | | | | | | | | | | |
| Verify eligibility in chart review or from Dr. Letter: • Medical history • Demographics | Х | | | | | | | | | | | |
| Randomization | X | | | | | | | | | | | |
| Baseline Questionnaires (Listed below with) | X | | | | | | | | | | | |
| Shipment of VR device and/or study documents | Х | | | | | | | | | | | |
| Technical onboarding call | | X | | | | | | | | | | |
| Milligram Morphine<br>Equivalent (MME) Daily Dose | X | | | | | | | | | Х | | |
| Return of VR Device | | | | | | | | | | | Х | |
| Deliver honorarium | | | | | | X | | | | Х | | X |
| | Se | If-Repo | rted | Questi | onnaire | es | | | | | | |
| NIH developed baseline demographics, biological sex | X (Day 1) | | | | | | | | | | | |
| Daily Pain Medications Used | Х | | | | | | | | | Х | | |
| Daily Pain Intensity | X | | | | | | | | | X | | |
| Pain Catastrophizing Scale | X (Day 4) | | Χ | Х | Х | Х | X | Х | Х | X | | |
| PROMIS Anxiety Scale | X (Day 4) | | Х | Х | Х | Х | Х | Х | Х | Х | | |
| PROMIS Pain Interference<br>Scale | X (Day 4) | | Х | Х | Х | Х | Х | Х | Х | Х | | |
| The Pain Self-Efficacy<br>Questionnaire (PSEQ) 2-item<br>short form | X (Day 4) | | х | Х | х | Х | Х | х | х | х | | |
| Simulator Sickness Questionnaire (VR only) | | X | | | | | | | | | | |
| Treatment Usage<br>Questionnaire | | | Х | Х | Х | Х | Х | Х | Х | Х | | Х |
| Events Assessment | | | Х | Х | Х | Х | Х | Х | X | Х | | |
| Custom Questions | | X | | | | | | | | Х | | |
| Treatment Expectation | X (Day 4) | Х | | | | | | | | | | |
| Concomitant Procedures Questionnaire | X (Day 4) | | | | | | | | | X | | |
| Primary Pain Questionnaire | | | | | | | | | | X | | |
| Coping with Weekly Pain<br>Questionnaire | X (Day 7) | | | | | | | | | X | | Х |